CLINICAL TRIAL: NCT04364828
Title: NGS Diagnostic in COVID-19 Hosts - Genetic Cause Relating to the Course of Disease Progression
Acronym: COVID-19 NGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: COVID-19 NGS
Record Dates: First submitted 2020-04-22; First posted 2020-04-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; Next-Generation-Sequencing; Whole Genome Analysis; MultiOmics; Extreme phenotypes
MeSH Terms: conditions — COVID-19 | interventions — Genome-Wide Association Study; Receptors, Antigen, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Host Genome Analysis (Other): For 150 patients from the extreme phenotypes - complementary to Whole Genome Analysis of each patient also Whole Transcriptome will performed Analysis; DNA methylation analysis using EPIC arrays will be performed in the pilot study (phase 1). Identically, in phase 2 starting from month 4, will be generated WGS, Whole transcriptome sequencing (WTS), and methylation data of the 500 patients. Epigenetic changes are likely to occur upon Corona infection. Subsequently, genome and epigenome data with RNA expression pattern will be correlated.
  Interventions: Genetic: Whole Genome Analysis
- Host Response to SARS-CoV-2 Infection (Other): Focus on longitudinal analysis of TCR repertoire of CD4+ and CD8+ T cells from blood samples (PBMCs) from clinically characterized patients (n = 24). The bulk- T-cell receptor (TCR) sequencing will be performed at different time points during the course of disease progression and recovery.
  Interventions: Genetic: T-cell receptor (TCR) repertoire
- Viral Sequence Composition (Other): The Severe Acute Respiratory Syndrome-Corona Virus-2 (SARS-CoV-2) viral composition is determined by Next Generation sequencing (different protocols for enrichment are available, and are currently being tested to successfully analyse the virus from different isolates). It is known that SARS-CoV-2 sequence is changing at least one position every second passing from person to person. Numerous variants have been described deriving from 3 different ancestral viruses (named A, B, and C) reflecting different distributions in East Asia, Europeans and Americans. At it is anticipated that other (super)infections may add to the severity of the infection and disease course, the entire metagenome of the throat is being sequenced and analyzed as well.
  Interventions: Genetic: SARS-CoV-2 viral composition

INTERVENTIONS:
Genetic: Whole Genome Analysis — Whole Genome Analysis with whole transcriptome analysis and deoxyribonucleic acid (DNA) methylation analysis using Methylation beadchip (EPIC) arrays
  Arms: Host Genome Analysis
Genetic: T-cell receptor (TCR) repertoire — Longitudinal analysis of TCR repertoire of Cluster of Differentiation 4+ (CD4+) and CD8+ T cells from blood samples (Peripheral Blood Mononuclear Cells, PBMCs) from clinically characterized patients
  Arms: Host Response to SARS-CoV-2 Infection
Genetic: SARS-CoV-2 viral composition — Determined by Next Generation sequencing
  Arms: Viral Sequence Composition

SUMMARY:
In this study (i) the host genome to identify susceptibility regions of infection, inflammation, and host defense, (ii) host response to Severe Acute Respiratory Syndrome-Corona-Virus-2 (SARS-CoV-2) infection, and (iii) viral sequence composition to define viral sequences which may be correlated with disease severity in addition to the metagenome of the throat swab will be analysed .

DETAILED DESCRIPTION:
This study aims to recruit adult persons with diagnostically confirmed Corona-Virus- Disease-19 (COVID-19) infection and with different disease manifestation who are included into diagnostic or therapeutic care at the University Hospital Tübingen (UKT).

The COVID-19 Next-Generation-Sequencing (NGS) study aims to cover as many patients in Germany as possible. It is expected to include in Phase 1 (pilot study): 250 patients with different disease manifestation (extreme phenotypes) and individual risk factors by whole genome analysis Phase 2 (verification study): 1.000 clinically well-defined patients to ensure a broader range of overlapping phenotypes, to verify data from the pilot study.

Phase 3 (confirmation study): > 10.000 patients to increase the power (anticipated).

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 infection confirmed
* COVID-19 disease manifestation
* Age > 18 years

Exclusion Criteria:

* Missing informed consent of the patient/ legal guardian/ relatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Viral evolution | Day 1, Day 3-5, Day 7-9, 48 hours after recovery
  The change in the genetic makeup of a virus population (measured in numbers) as the viruses mutate and multiply over time at different time points

SECONDARY OUTCOMES:
Immune response | Day 1, Day 3-5, Day 7-9, 48 hours after recovery
  CD4+ and CD8+ T cells from blood (per µl) at different time points measured
Disease severity | Day 1, Day 3-5, Day 7-9, 48 hours after recovery
  Clinical classification according to severity:
  * Light and uncomplicated (mild symptoms)
  * Moderate (mild pneumonia)
  * Severe pneumonia
  * Critical (Acute Respiratory Distress Syndrome (ARDS), sepsis, septic shock) Evaluated at several time points

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Rieß, Prof. Dr., Study Director — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Yes
The COVID-19 NGS study will provide data in a pseudonymized manner to national and international databases set up to increase the diagnostic yield through advanced analysis tools.
Supporting Information: Analytic Code
Time Frame: Data will become available after analysis and unlimited.
Access Criteria: Authorized users within the participating organizations.